CLINICAL TRIAL: NCT04562831
Title: A Randomized Placebo-controlled Trial of Nicotinamide/Pterostilbene Supplement in ALS: The NO-ALS Study
Brief Title: The NO-ALS Study: A Trial of Nicotinamide/Pterostilbene Supplement in ALS.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Elysium Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 98955
Record Dates: First submitted 2020-09-10; First posted 2020-09-24 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — nicotinamide-beta-riboside; Pterocarpus marsupium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Newly diagnosed ALS patients (Experimental): 1. High dose EH301 (1500mg Nicotinamide riboside / 300mg Pterostilbene)
  2. Single dose EH301 (1000mg Nicotinamide riboside / 200mg Pterostilbene)
  3. Placebo
  Interventions: Dietary Supplement: EH301 (Nicotinamide Riboside/Pterostilbene)
- Earlier diagnosed ALS patients (Experimental): 1. High dose EH301 (1500mg Nicotinamide riboside / 300mg Pterostilbene)
  2. Placebo
  Interventions: Dietary Supplement: EH301 (Nicotinamide Riboside/Pterostilbene)

INTERVENTIONS:
Dietary Supplement: EH301 (Nicotinamide Riboside/Pterostilbene) — Comparison of 2 different dosages with placebo in newly diagnosed ALS patients and comparison of high dose with placebo in earlier ALS patients.

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a serious rapidly progressive disease of the nervous system. The average survival from the time of diagnosis is 3 years. Apart from Riluzole, there is no effective treatment. Care of advanced ALS will have a cost of 4-8 million NOK per year

Research i.a. from the investigators department has shown that increased activity in histone deacetylation enzymes (sirtuins) together with increased access to NAD can delay disease progression. Nicotinamide riboside (NR) can increase cells' access to NAD and Pterostilben will stimulate sirtuins.

The investigators want to study whether combination therapy with NR and Pterostilben can inhibit neurodegeneration in ALS and thereby delay disease development, increase survival and improve quality of life in ALS.

In the study, the investigators will use 2 different dosages on the active treatment and strength calculations show that 180 patients are needed to show a rather weak effect. Patients will be recruited in collaboration with hospitals in Helse Vest, AHUS, Drammen, OUS and St. Olavs hospital.

ELIGIBILITY:
Inclusion Criteria:

Arm 1 (newly diagnosed ALS patients)

* Have a clinical diagnosis of probable ALS according to the revised El Escorial criteria.
* MR of the brain and cervical spine cannot explain symptoms.
* Diagnosed with likely ALS within 6 months from enrolment and treated with Riluzole 50mg x 2
* Symptom onset no longer than 2 year prior to inclusion.
* ALS-FRC-R of 36 or more (not any item below 2).
* Age equal to or greater than 35 years at time of enrollment

Arm 2 (earlier diagnosed ALS patients)

* Have a clinical diagnosis of probable ALS according to the revised El Escorial criteria.
* MR of the brain and cervical spine cannot explain symptoms.
* Treated with Riluzole 50mg x 2.

Exclusion Criteria:

* Dementia, FTD or other neurodegenerative disorder at baseline visit
* Any psychiatric disorder that would interfere with compliance in the study.
* Use of high dose vitamin B3 supplementation within 30 days of enrollment
* Metabolic, neoplastic, or other physically or mentally debilitating disorder at baseline visit.
* Genetically confirmed mitochondrial disease
* Patients who become tracheostomized as part of the treatment of ALS
* Patients with short expected survival at the discretion of the investigator. Such cases cannot be expected to follow protocol procedures.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2020-10-07 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Disease progression as assessed by Amyotrophic Lateral Sclerosis Functional Rating Scale Revised (ALSFRS-R) | Change from baseline to 1 year
  ALSFRS-R is a validated rating instrument for monitoring the progression of disability in patients with ALS. The minimum score is 0 and the maximum score is 48, the higher score the more function is retained.

SECONDARY OUTCOMES:
Change in vital capacity | Change from baseline to 1 year
  Vital capacity in sitting position and supine by spirometry. Spirometry measures the amount of air that can be inhaled or exhaled and vital capacity is the volume of air breathed out after the deepest inhalation, the higher value the better vital capacity.
Change in cognitive functions as assessed by the Edinburgh Cognitive Scale (ECAS) | Change from baseline to 1 year
  ECAS determines cognitive and behavioural changes of patients suffering from ALS. The minimum score is 0 and the maximum score is 136, the lower the score the greater the deficit.
Change of Neurofilament light chain (NFL) levels in serum | Change from baseline to 1 year
  NFL levels in serum, baseline values and changes during the study.
Change in quality of life as assessed by the quality of life questionnaire SF-36 | Change from baseline to 1 year
  SF-36 is a 36-item patient-reported survey of patient health. The minimum score is 0 and the maximum score is 100. The higher the score the less disability.

OTHER OUTCOMES:
Overall survival | Through study completion, 1 year
  Survival of patients through the study

CONTACTS AND LOCATIONS:
Overall Officials: Ole-Bjørn Tysnes, Principal Investigator — Haukeland University Hospital
Locations (9):
- Norway (9):
  - Haukeland University Hospital, Bergen
  - Vestre Viken HF, Drammen
  - Helse Førde HF, Førde
  - Helse Fonna HF, Haugesund
  - Akershus University Hospital, Lørenskog
  - Oslo University Hospital, Oslo
  - Stavanger University Hospital, Stavanger
  - Universitetssykehuset Nord-Norge, Tromsø
  - St.Olavs Hospital HF, Trondheim

IPD SHARING:
Plan to Share IPD: No